CLINICAL TRIAL: NCT05375110
Title: A Prospective, Multi-center and Objective Performance Criteria Study to Evaluate the Effectiveness and Safety of NoYA™ Radiofrequency Interatrial Shunt System for the Treatment of Chronic Heart Failure With Elevated Left Atrial Pressure
Brief Title: NoYA RAISE Trial II (Radiofrequency Ablation-Based Interatrial Shunt for Heart Failure)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou NOYA MedTech Co. Ltm. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOYA-01
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Heart Failure with Preserved Ejection Fraction [HFpEF]; Heart Failure with Reduced Ejection Fraction [HFrEF]
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NoYA™ Radiofrequency Interatrial Shunt System (Experimental): Eligible patients will be enrolled and undergo radiofrequency ablation of the interatrial procedure with the NoYA™ Radiofrequency Interatrial Shunt System (Noya Medtech).
  Interventions: Device: NoYA™ Radiofrequency Interatrial Shunt System

INTERVENTIONS:
Device: NoYA™ Radiofrequency Interatrial Shunt System — NoYA™ Radiofrequency Interatrial Shunt System include Adjustable Interatrial Shunt System and Radiofrequency Ablation Generator.

SUMMARY:
A Prospective, Multiple Center, and Objective Performance Criteria Study to Evaluate the NoYA™ Radiofrequency Interatrial Shunt System manufactured by NoYA Medtech (Hangzhou) Co., Ltd. for the Treatment of Chronic Heart Failure with Elevated Left Atrial Pressure.

DETAILED DESCRIPTION:
This is a prospective, multi-center and objective performance criteria study to evaluate the effectiveness and safety of the NoYA™ Radiofrequency Interatrial Shunt System for the treatment of chronic heart failure with elevated left atrial pressure. Patients with chronic heart failure with elevated left atrial pressure who meet study eligibility criteria will be enrolled and undergo radiofrequency ablation of the interatrial procedure with NoYA™ Radiofrequency Interatrial Shunt System (Noya Medtech) after signing the informed consent. The follow-up will be conducted at discharge, 1 month, 3 months, 6 months, and 12 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. Chronic symptomatic Heart Failure (HF) documented by one or more of the following:

   1. New York Heart Association (NYHA) Class II/III/ambulatory class IV symptoms (Paroxysmal nocturnal dyspnea, Orthopnea, Dyspnea on mild or moderate exertion) at screening visit; or signs (Any rales post cough, Chest x-ray demonstrating pulmonary congestion,) within past 12 months;
   2. One hospital admission for which HF was a major component of the hospitalization within the 12 months prior to study entry (transient heart failure in the context of myocardial infarction does not qualify).
3. Sustained and stable GDMT (guideline-directed medical therapy) for heart failure according to the 2017 ACC/AHA/HFSA guidelines management as well as potential complications of heart failure management, heart failure symptoms remain uncontrolled.
4. LV ejection fraction (EF) ≥15% measured by echocardiography in the last 6 months.
5. Invasive hemodynamic measurements showed mLAP or end-expiratory resting PCWP≥15mmHg, and mLAP or PCWP-RAP ≥5mmHg.
6. Subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, as approved by the IRB.

Exclusion Criteria:

1. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
2. Bacterial endocarditis.
3. 6-minute walk test distance <100m or > 450m.
4. History of atrial septum implantation (e.g. atrial septum occlusion, patent foramen ovale occlusion) or inferior vena cava filter.
5. History of myocardial infarction (MI), percutaneous coronary intervention (PCI), or coronary artery bypass grafting (CABG) within the past 3 months; Untreated severe coronary artery stenosis which requires revascularization.
6. History of cardiac resynchronization therapy (CRT/CRT-D) or implantable cardioverter-defibrillator (ICD) implantation within the past 6 months.
7. Right heart failure
8. Pulmonary arterial hypertension (TTE or cardiac catheterization shows pulmonary artery systolic pressure>70mmHg)
9. Life expectancy less than 12 months.
10. In the opinion of the investigator, the subject is not an appropriate candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of free from death and heart failure (HF) related hospitalizations at 12 months follow-up | 12 months after the procedure
  1. Death: Cardiac death
  2. Hospitalization：HF-related Hospitalizations

SECONDARY OUTCOMES:
Acute device success | Immediately post-procedure
  Acute device success is defined as the successful delivery and retraction of the device without immediate postoperative device-related technical failures or complications.
Acute procedural success | Immediately post-procedure
  Acute procedural success is defined as no operative death immediately after the operation, successful delivery and fully retraction of the device, no need for any emergency surgery or secondary intervention (including device-related or operative approach-related), and the presence of the left-to-right atrial blood shunt (means the shunt is patent).
Change in 6-Minute Walk Test | Baseline, 6 months, 12 months after procedure
  The change of 6-minute walk test distance between baseline, 6 months, and 12 months follow-up.
Change in Nt-pro BNP | Preoperative, 1 month, 3 months, 6 months, 12 months after procedure
  Change in Nt-pro BNP between preoperative, 1 month, 3 months, 6 months, and 12 months follow-up.
Change in PCWP or Mean Left Atrial Pressure | Before, immediately after procedure
  Change in resting end-expiratory PCWP (pulmonary capillary wedge pressure) or mean left atrial pressure before and immediately after the procedure.
Left-to-right Atrial Blood Shunt Evaluation | 6 months, 12 months after procedure
  Echocardiographic assessment of left-to-right atrial blood shunt at 6 months and 12 months postoperatively: peak shunt flow rate, maximum shunt orifice diameter.
Change in NYHA Class | Preoperative, 1 month, 3 months, 6 months, 12 months after procedure
  Preoperative, 1 month, 3 months, 6 months, and 12 months postoperative cardiac function class (NYHA class).
Change in Minnesota Living with Heart Failure Questionnaire | Preoperative, 1 month, 3 months, 6 months, 12 months after procedure
  Preoperative, 1 month, 3months, 6 months, and 12 months postoperative Quality of life assessment in Minnesota Living with Heart Failure Questionnaire.
Rate of re-admission, re-operation/intervention for heart failure | 12 months after procedure
  The overall incidence of re-admission, re-operation/intervention for heart failure within 1 year.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Hainan General Hospital, Hainan, Hainan
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The 7th People Hospital of Zhengzhou, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Yantai YuHuangDin Hospital, Yantai, Shandong
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The Shanghai Ninth People's Hospital affiliated with the Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No